CLINICAL TRIAL: NCT05135975
Title: Phase 2 Study of Cabozantinib as a Maintenance Agent to Prevent Progression or Recurrence in High-Risk Pediatric Solid Tumors
Brief Title: A Study of Cabozantinib as a Maintenance Agent to Prevent Progression or Recurrence in High-Risk Pediatric Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CaboMain
Record Dates: First submitted 2021-11-04; First posted 2021-11-26 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Neuroblastoma; Sarcoma
Keywords: Malignant rhabdoid tumor; Osteosarcoma; Ewing sarcoma; Rhabdomyosarcoma; Desmoplastic small round blue cell tumor; Wilms tumor; Solid tumor; Metastatic osteosarcoma
MeSH Terms: conditions — Neuroblastoma; Sarcoma; Rhabdoid Tumor; Osteosarcoma; Sarcoma, Ewing; Rhabdomyosarcoma; Wilms Tumor | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cabozantinib (Experimental): Enrolled patients will be treated with cabozantinib maleate, tablet formulation, using the recommended Phase 2 dose of 40 mg/m2/day, to a maximum of 420 mg/week. Treatment will be administered in 28- day cycles.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Enrolled patients will be treated with cabozantinib maleate, tablet formulation, using the recommended Phase 2 dose of 40 mg/m2/day to a maximum of 420 mg/week. Treatment will be administered in 28- day cycles.

SUMMARY:
This study will expand the types of pediatric cancers being evaluated for response to cabozantinib. The current COG study is restricted to Ewing sarcoma, osteosarcoma, rhabdomyosarcoma, Wilms tumor, and a handful of uncommon tumors. The proposed study will extend this evaluation to tumors that have been shown to either express known targets of cabozantinib or with preclinical evidence of efficacy, including specifically neuroblastomas. These tumors have high morbidity and mortality, particularly in the relapse setting, and few or no proven therapeutic options. As such, evaluation of cabozantinib in these studies is warranted.

The study hypothesizes that use of cabozantinib in patients with ultra-high-risk pediatric solid tumors with minimal disease burden, as defined in the inclusion criteria below, can prevent and/or slow recurrent tumor formation in pediatric solid tumors and thereby significantly extend the period of disease control and/or induce a durable cure.

DETAILED DESCRIPTION:
The study hypothesizes that use of cabozantinib in patients with ultra-high-risk pediatric solid tumors who have achieved and maintained (for at least 4 weeks) a "best response" to their most recent line of therapy, as defined in the inclusion criteria below, can prevent and/or slow recurrent tumor formation in pediatric solid tumors, improve one-year progression-free survival by 20% as compared to historical controls, and also improve longer-term progression-free and overall survival without significant impact on quality of life. We also hypothesize, in an exploratory aim, that there will be improvement in two-year progression free survival in patients with metastatic Ewing sarcoma and osteosarcoma specifically.

The study proposes to evaluate the efficacy of up to one year of treatment with cabozantinib in pediatric solid tumors after completion of last therapy with a "best response." There are multiple reasons for this approach, as opposed to continual therapy until toxicity or disease progression alone. First, for most of these ultra-high-risk diseases, the greatest risk of recurrence has historically been within 12 months after last therapy, and often times considerably sooner. As such, we should be able to evaluate a meaningful difference within 12 months. Second, the goal of this study is to evaluate if, during a critical period of disease control, use of cabozantinib can induce a durable remission. There are active Phase 2 and 3 studies of cabozantinib, including with the Children's Oncology Group, evaluating the efficacy of cabozantinib in controlling pediatric cancers with measurable burden of disease. However, we know that, in patients with "ultra-high-risk" disease who have achieved a best response including stable disease, partial response or even complete response, there is still active disease with high risk of growth, as demonstrated in the studies cited above. Our study seeks to augment ongoing work in pediatric cancers by testing the hypothesis that cabozantinib can durably silence cancer cell viability after a best response to prior treatment. Third, this work would mark a fundamental change in the indication for use of cabozantinib in pediatric cancers, broadening its utility from a "rescue" agent to a maintenance therapy that may be critical for disease control, during either primary or secondary remission.

This study will expand the types of pediatric cancers being evaluated for response to cabozantinib. The current COG study is restricted to Ewing sarcoma, osteosarcoma, rhabdomyosarcoma, Wilms tumor, and a handful of uncommon tumors. The proposed study will extend this evaluation to tumors that have been shown to either express known targets of cabozantinib or with preclinical evidence of efficacy, including specifically neuroblastomas. These tumors have high morbidity and mortality, particularly in the relapse setting, and few or no proven therapeutic options. As such, evaluation of cabozantinib in these studies is warranted.

ELIGIBILITY:
3.2 Patient Eligibility Criteria:

3.2.1 Assessment criteria for eligibility, based on disease burden at start of most recent line of therapy and corresponding response (patients must meet one of the following criteria in order to be deemed eligible for enrollment):

1. Patients previously with measurable disease, at start of most recent line of therapy, AND without evaluable disease (or for whom assessment of potential evaluable-only disease would not be considered standard of care) are eligible based on "measurable disease response" only in Section 3.1.2.a.i.
2. Patients previously with evaluable disease at start of most recent line of therapy, AND without measurable disease at that time are eligible based on "evaluable disease" definition alone only in Section 3.1.2.a.ii.
3. Patients previously with measurable AND evaluable disease at start of most recent line of therapy must meet BOTH "measurable disease" and "evaluable disease" definitions under Section 3.1.2.a.

3.2.2. Disease Strata. Patients need to meet any single definition of disease below:

1. Stratum A: Solid tumors with 1-year PFS ≤25% (target enrollment 36 patients)

   1. Neuroblastoma BR1 at the end of frontline therapy with residual disease (less than complete response (CR), including MIBG-avid stable disease as per Section 3.1.2.a.ii,.or >5% bone marrow involvement) but not progressive at time of enrollment
   2. Neuroblastoma BR2 or later.
   3. Osteosarcoma, BR2 or later
   4. Ewing sarcoma, BR2 or later
   5. Rhabdomyosarcoma, with positive surgical margins OR with primary extremity tumor with >2 metastases at diagnosis, BR1 or later
   6. Rhabdomyosarcoma, alveolar subtype or fusion-positive subtype, BR2 or later
   7. Rhabdomyosarcoma, embryonal subtype, Group 4 at original diagnosis, BR2 or later
   8. Desmoplastic small round blue cell tumor, BR2 or later
   9. Any other soft tissue sarcoma, BR2 or later
   10. Wilms tumor, diffuse anaplasia histology, any stage, BR2 or later
   11. Wilms tumor, any histology with relapse within 12 months of diagnosis, who have received prior treatment with doxorubicin, and intraabdominal recurrence, BR2 or later
   12. Wilms tumor, BR3 or later
   13. Other solid tumor with 1-year PFS ≤ 20% can be discussed with study chair for eligibility
2. Stratum B: Metastatic Ewing sarcoma with metastases not undergoing complete metastatectomy, BR1 (target enrollment 20 patients)
3. Stratum C: Metastatic osteosarcoma after frontline therapy, BR1 (target enrollment 20 patients)
4. Stratum D: Metastatic fusion-positive rhabdomyosarcoma after frontline therapy, BR1 (target enrollment 10 patients)

3.2.3 Inclusion Criteria for Eligibility:

1. Age: ≥ 18 months of age and <40 years of age at time of study enrollment
2. Performance level: Patients must have a Lansky or Karnofsky performance status score of ≥ 50, corresponding to ECOG categories 0, 1 or 2. Use Karnofsky for patients > 16 years of age and Lansky for patients ≤ 16 years of age. Patients who are unable to walk because of paralysis, but who are upright in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score. Patients should also have recovery to baseline or ≤ Grade 1 CTCAE v4.03 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy (see Section 3.2.3, criteria 4)
3. Patient Body Surface Area (BSA): Patients must be ≥0.35 m2 in BSA, using the Mosteller formula, BSA = (((Height in cm) * (Weight in kg))/ 3600)½ within two weeks of study enrollment
4. Prior therapy: patients must have recovered from the acute toxic effects of prior therapy, with the following time specifications:

   1. Myelosuppressive chemotherapy: Patients must not have received myelosuppressive chemotherapy within 3 weeks of enrollment on study (6 weeks if prior therapy included nitrosourea)
   2. Other medicinal anti-cancer agents: Patients must not have received non-myelosuppressive anticancer agents, including any type of small molecule kinase inhibitor, within 14 days of enrollment on study
   3. Biological anticancer therapy (including antibody therapy or cellular therapy): Patients must not have received biological anticancer therapy within 21 days of enrollment on study
   4. Radiation therapy: Patients must not have received external beam radiation therapy to sites outside of the lungs within 2 weeks of study enrollment, external beam radiation therapy to sites within the lungs within 4 weeks of study enrollment, or I-131 MIBG therapy within 6 weeks of study enrollment. Subjects with clinically relevant ongoing complications from prior radiation therapy MUST be discussed with Study Chair or his proxy to determine suitability and safety of enrollment.
   5. Myeloablative therapy: Patients must not have received myeloablative therapy within 2 months of study enrollment, must not have received a blood stem cell/marrow infusion within 3 weeks of study enrollment, and must have attained blood count recovery as per Section 3.2.3, criteria 5
5. Bone Marrow Function: Patients must have adequate bone marrow function at time of study enrollment, as defined as:

   1. Absolute neutrophil count (ANC) ≥1000/mcL; patients cannot have received filgrastim, pegfilgrastim or equivalent biosimilar within 14 days of study enrollment
   2. Platelet count ≥ 100,000/mcL; patients can receive no more than 15 mL/kg of platelet transfusions per week at time of enrollment to meet the parameters; patients can receive a TPO agonist (e.g., eltrombopag or romiplostim) at time of enrollment but must be on a stable dose for at least 14 days prior to enrollment
   3. Hemoglobin ≥ 8.0 g/dL; patients can receive no more than 10 mL/kg of packed red blood cells (PRBCs)/week transfused at time of enrollment on therapy to meet the parameters; patients may receive erythropoietin or biosimilar equivalent but must have been on a stable dose and not require PRBC transfusions for at least 14 days prior to study enrollment
   4. Patients with residual bone marrow metastases at end of most recent line of therapy must have stable disease or better at two bone marrow evaluations at least 4 weeks apart, with the second marrow assessment at least 4 weeks after end of most recent therapy. Stable disease is defined as <2-fold change in marrow burden between the two timepoints and ≤20% marrow involvement. When bilateral bone marrow assessment is performed, average marrow involvement of the two sites will be used for eligibility.
6. Renal Function: Patient must meet criteria for both a. and b. below to have adequate renal function, within 2 weeks of study enrollment

   1. Creatinine clearance or radioisotope GFR ≥ 70 mL/min/1.73 m2, as per institutional standard testing OR serum creatinine based on age/gender as listed in protocol:
   2. Urine protein: ≤ 30 mg/dl in urinalysis (clean catch recommended), equivalent to ≤ 1+ on dipstick OR quantitative urine protein < 1000 mg in a 24hr urine sample. NOTE: If the initial urinalysis shows >30 mg/dL urine protein (or > 1+ on dipstick), a 24-hour quantitative urine protein should be utilized, as described above, for eligibility consideration.
7. Hepatic function: Patient must meet ALL of the below criteria, within 14 days of study enrollment, to have adequate hepatic function:

   1. Total bilirubin < 2x institutional upper limit of normal (ULN) for age
   2. ALT<5x ULN
   3. Serum albumin >2.7 g/dL
8. Cardiovascular Function: Patients must have adequate cardiovascular function as defined as:

   1. No significant arrhythmias, strokes, transient ischemic attacks, or myocardial infarction within 6 months of study enrollment
   2. QTc ≤ 480 msec within 7 days of study enrollment (calculated using Bazett calculation or Fridericia calculation as per institutional standard of care; whichever calculation is used for eligibility must be used for all future QTc calculations).

      A single ECG with QTc meeting the above criterion is adequate. However, if an initial ECG shows a QTc >480 ms, obtain two additional ECGs with each ECG at least 30 minutes apart. Calculate each individual QTc by the same calculation method and average the values; the resulting average QTc will be used for eligibility.
   3. Blood pressure ≤ 95th percentile for age, height, and gender for patients <18 years of age (78), or BP ≤140/90 for patients ≥18 years of age. At time of enrollment, patients may be on one antihypertensive agent at a stable dose for at least 2 weeks prior to enrollment.
9. Pancreatic function: Patient must have adequate pancreatic function, as defined by a serum lipase <2x ULN
10. Neurologic function: Patients with defined seizures who are on a stable anti- convulsant regimen using drugs that do not induce hepatic metabolizing enzymes for at least 4 weeks are eligible for enrollment Recommended Non-enzyme inducing anticonvulsants Clonazepam Diazepam Ethosuximide Ezogabine Gabapentin Lacosamide Lamotrigine Levetiracetam Lorazepam Perampanel Tiagabine Topiramate Valproic Acid Zonisamide Unacceptable Enzyme inducing anticonvulsants Carbamazepine Felbamate Phenobarbital Fosphenytoin Phenytoin Primidone Oxcarbazepine
11. Lung integrity: Patients must not have had any invasive pulmonary procedure (including bronchoalveolar lavage, lung biopsy, transbronchial biopsy, or thoracotomy) or pneumothorax within 4 weeks of enrollment on study.
12. Surgeries or trauma:

    1. Patients must not have had any major surgical procedures, laparoscopic procedures, sepsis, shock, or physical trauma requiring hospitalization within 4 weeks of enrollment on study. The primary surgeon of any major surgical procedures must authorize antineoplastic treatment before enrollment on study.
    2. Patients must not have had a central line or subcutaneous port placement, revision, or removal (excluding a peripherally inserted central catheter (PICC)) within 7 days of study enrollment. Advise patients with a surgically placed central line or subcutaneous port that removal of the port once enrolled on study would require holding study treatment for 4 weeks prior, and surgical removal of the central line or port would be recommended to be performed prior to cabozantinib initiation.
    3. Patients must not have had a core or fine needle biopsy within 7 days of study enrollment.
    4. Any surgical wounds or incisions must be healed, as determined by treating physician, prior to enrollment on study.
    5. Bone marrow aspiration and/or biopsy are not considered surgical procedures for the purpose of this study.
13. Patients must be able to swallow tablets intact. Tablets cannot be cut or crushed.
14. Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (eg, barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 4 months after the last dose of study treatment. Post-menarchal females must be confirmed to not be pregnant at time of enrollment.
15. Patient or legal guardian must be capable of understanding and complying with the protocol requirements and must have signed the informed consent document.
16. Patient must be able to start study treatment no later than 12 weeks after end of prior therapy, where 1 week = 7 days.
17. Patient must be enrolled on study within 14 days of qualifying radiographic imaging studies demonstrating best response as per Section 3.1.2.
18. Patient must be able to start study treatment no later than 7 days from study enrollment.

SEE PROTOCOL FOR ADDITIONAL EXCLUSION CRITERIA

Ages: 18 Months to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of oral daily cabozantinib, administered for up to 12 months, on the one-year progression-free survival of patients with "ultra-high-risk" pediatric solid tumors. | 4 years
  Defined as the time from diagnosis until the date of disease progression

SECONDARY OUTCOMES:
To evaluate the effect of oral daily cabozantinib on the one-, two-, and five-year overall survival of patients with "ultra-high-risk" pediatric solid tumors. | 5-8 years
  Defined as the time from initiation of therapy to the date of death
To evaluate the effect of oral daily cabozantinib on the two- and five-year progression- free survival of patients with "ultra-high-risk" pediatric solid tumors. | 8 years
  Defined as the time from diagnosis until the date of disease progression
To evaluate the duration of response to cabozantinib, both during drug administration and after discontinuation of cabozantinib at study-defined time points. | 4 years
  Response rate = occurrence of partial response (PR) or complete response (CR)
To evaluate the incidence of adverse events associated with the use of cabozantinib in this population when taken for up to 12 months. | 4 years
  Adverse events will be defined using the CTCAE v.4.03

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Shah, MD, Principal Investigator — Nationwide Children's Hospital
Locations (6):
- United States (6):
  - Children's Hospital of Alabama/UAB, Birmingham, Alabama
  - Children's Hospital of Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Hospital at Montefiore, The Bronx, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Primary Children's Hospital, Salt Lake City, Utah